CLINICAL TRIAL: NCT06935266
Title: A Phase 1, Open-Label, Within-Dose-Level Randomized Trial to Assess the Tolerability, Safety, and Pharmacokinetics of Immune Globulin Subcutaneous 20% (Human) With Recombinant Human Hyaluronidase (TAK-881) With Ramp-Up and No Ramp-Up Dosing in Healthy Adult Participants
Brief Title: A Study of TAK-881 With and Without Ramp-Up Dosing in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-881-1003
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (8):
- Cohort 1, Schedule B, Treatment Arm 1: TAK-881 (Experimental): Participants will receive TAK-881, subcutaneous (SC) injection, 0.15 grams per kilogram (g/kg) on Day 1, 0.3 g/kg on Day 8, 0.6 g/kg on Days 22 and 50 in ramp-up dosing manner.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets
- Cohort 1, Schedule C, Treatment Arm 2: TAK-881 (Experimental): Participants will receive TAK-881, SC injection, 0.6 g/kg on Days 1, 29 and 57 in no ramp-up dosing manner.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets
- Cohort 2, Schedule A, Treatment Arm 3: TAK-881 (Experimental): Participants will receive TAK-881, SC injection, 0.25 g/kg on Days 1 and 8, 0.5 g/kg on Day 15, 0.75 g/kg on Day 29 and 1.0 g/kg on Day 50 in ramp-up dosing manner.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets
- Cohort 2, Schedule B: Treatment Arm 4: TAK-881 (Experimental): Participants will receive TAK-881, SC injection, 0.25 g/kg on Day 1, 0.5 g/kg on Day 8, 1.0 g/kg on Days 22 and 50 in ramp-up dosing manner.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets
- Cohort 2, Schedule C: Treatment Arm 5: TAK-881 (Experimental): Participants will receive TAK-881, SC injection, 1.0 g/kg on Days 1, 29 and 57 in no ramp-up dosing manner.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets
- Cohort 3, Schedule A: Treatment Arm 6: TAK-881 (Experimental): Participants will receive TAK-881, SC injection, 0.5 g/kg on Days 1 and 8, 1.0 g/kg on Day 15, 1.5 g/kg on Day 29 and 2.0 g/kg on Day 50 in ramp-up dosing manner.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets
- Cohort 3, Schedule B: Treatment Arm 7: TAK-881 (Experimental): Participants will receive TAK-881, SC injection, 0.5 g/kg on Day 1, 1.0 g/kg on Day 8, 2.0 g/kg on Days 22 and 50 in ramp-up dosing manner.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets
- Cohort 3, Schedule C: Treatment Arm 8: TAK-881 (Experimental): Participants will receive TAK-881, SC injection, 2.0 g/kg, on Days 1, 29 and 57 in no ramp-up dosing manner.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets

INTERVENTIONS:
Biological: TAK-881 — TAK-881 SC injection.
  Other Names: Immune Globulin Subcutaneous (Human), 20% Solution with Recombinant Human Hyaluronidase (rHuPH20); 20% Solution with Recombinant Human Hyaluronidase (rHuPH20)
Device: SC Investigational Needle Sets — The single-use only SC needle set will be used to administer TAK-881 to the target depth below the skin surface. One needle set (single or bifurcated) will be used per infusion.

SUMMARY:
The main aim of this study is to check how well healthy adults can tolerate TAK-881 with different dosing schedules.

During the study, participants will receive one infusion of TAK-881 under the skin (subcutaneous [SC] infusion) on Day 1 at a lower dose level followed by participants receiving multiple infusion of higher dose levels.

Participants will be in the study for approximately 19 weeks including screening period and follow-up (End of Treatment [EOT]).

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women between 18 and 50 years can participate.
2. Must be a non-smoker, with no use of nicotine or tobacco products for at least 3 months prior to the first dosing.
3. Must have Body Mass Index (BMI) between 18.0 and 30.0 kilograms per square meter (kg/m^2).
4. Must be medically healthy.
5. Must follow protocol-specified contraception guidance.

Exclusion Criteria:

1. Any current or past medical history of blood/clotting disorder, liver, lung, heart, kidney, immune, skin, or brain or psychiatric condition.
2. History of alcohol or drug abuse within 2 years before dosing.
3. History or presence of hypersensitivity or severe allergic reactions to blood or blood components.
4. History or presence of thrombotic/thromboembolic events, or venous thrombosis.
5. Pregnant or breastfeeding.
6. Unable to refrain from taking prescription and non-prescription medications, herbal remedies, homeopathic preparations, or vitamin supplements.
7. Recently donated blood or blood products.
8. Participated in another clinical trial involving immunoglobulin products within 12 months of screening.
9. Has taken biologic agents within 12 weeks of screening.
10. Has used an investigational product within 30 days or 5 half-lives, whichever is longer, prior to screening.
11. Has received any vaccine (including live attenuated vaccines and coronavirus disease 2019 [COVID-19] vaccines) during the last 30 days before dosing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Tolerable Infusions of TAK-881 | From start of the study drug administration up to Day 57
  A tolerable infusion is considered to have occurred if an infusion is completed without interruption (discontinuing the infusion, or infusion rate reduction) due to any treatment-emergent adverse events (TEAEs) related to TAK-881.
Number of Tolerable Infusions | From start of the study drug administration up to Day 57
  A tolerable infusion is considered to have occurred if an infusion is completed without interruption (discontinuing the infusion, or infusion rate reduction) due to any TEAEs related to TAK-881.

SECONDARY OUTCOMES:
Number of Participants With TEAEs | From start of the study drug administration up to Week 16
  TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product.
Number of Participants With Clinically Significant Changes in Clinical Laboratory Values | Up to Week 16
  Laboratory parameters will include serum chemistry, hematology, coagulation and urinalysis. Clinical significance of laboratory values will be determined at the investigator's discretion.
Number of Participants With Clinically Significant Changes in Vital Sign Values | Up to Week 16
  Vital signs will include measurement of heart rate/ pulse rate, systolic, diastolic blood pressure, body temperature and respiratory rate. Clinical significance of vital signs will be determined at the investigator's discretion.
Number of Participants With Positive Binding Antibodies (Titer Greater Than or Equal to [>=] 1:160) | Up to Week 16
Number of Participants With Neutralizing Antibodies to rHuPH20 | Up to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/a3de9aa1c0df4e72